CLINICAL TRIAL: NCT01458431
Title: Efficacy of Continuous Infusion of Levobupivacaine to the Surgical Wound Following Cesarean
Brief Title: Levobupivacaine to the Surgical Wound Following Cesarean
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Manuel Ángel Gómez-Ríos (Other)
Responsible Party: Sponsor-Investigator, Manuel Ángel Gómez-Ríos, Principal Investigator, Complexo Hospitalario Universitario de A Coruña
Organization: Complexo Hospitalario Universitario de A Coruña (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGR-LB-2010-01
Record Dates: First submitted 2011-10-17; First posted 2011-10-24 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2011-10

CONDITIONS: Postoperative Pain
Keywords: cesarean section; wound infusion; Local anesthetic levobupivacaine; Pain management
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Levobupivacaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levobupivacaine (Experimental): Continuous levobupivacaine subfascial infusion
  Interventions: Drug: Levobupivacaine
- NaCl (Placebo Comparator): Continuous NaCl subfascial infusion
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Levobupivacaine — continuous levobupivacaine subfascial infusion
  Other Names: local anesthetic
  Arms: Levobupivacaine
Drug: NaCl — continuous NaCl subfascial infusion
  Other Names: Placebo
  Arms: NaCl

SUMMARY:
The postoperative period following cesarean is associated with moderate to severe pain that requires a considerable amount of analgesics that carry with them side-effects such as nausea, vomiting, fatigue and immobilization. Several studies have tried, with variable results, to find a more effective analgesia alternative such as infusion of local anesthetics through a catheter in the surgical wound sinus, a practice that has currently been widely used in clinical practice. Despite existing references on its use in the postoperative period following cesareans there continues to be a lack of information on other aspects. The investigators study hypothesis is that the use of levobupivacaine in the surgical wound will reduce the surface of hyperalgesia compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Full-term pregnant women who undergo scheduled cesarean surgery under intradural anesthesia.
* Duly informed patients who have signed the informed consent during the preanesthesia consultation, or after a period of consideration if necessary, expressing their consent to be included in the study.
* Between 18-45 years of age.
* ASA I and II.
* Sufficient intellectual ability to understand the technique as well as the equipment being used.

Exclusion Criteria:

* Failure to meet any of the above criteria.
* Presence of a major medical, cardiovascular, pulmonary, metabolic, renal or liver disorder.
* Preeclampsia and/or HELLP syndrome.
* Coagulopathy
* Profuse bleeding greater than 1000 ml or that which provokes hemodynamic instability that requires aggressive fluid therapy and/or transfusion.
* Allergy to any drug included in the protocol.
* Psychiatric or neurological pathology.
* Preexisting infection.
* Previous treatment with opioids or antidepressants or suffer from chronic pain.
* History of alcohol or drug abuse or known consumption of medications that interfere with LB metabolism.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2011-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area of incisional secondary hyperalgesia | 72 hours

SECONDARY OUTCOMES:
Pain relief | 72 hours
consumption of morphine (mg) and paracetamol (gr) | 48 hours
Incidence of chronic pain | 6 month
Pharmacokinetic variables of levobupivacaine | 72 hours
  Cmax, Area Under Curve, Tmax
Incidence of complications and/or side effects related to the technique | 72 hours
Rate of satisfaction experienced by the patients through a survey | 72 hours
endocrin-metabolic response | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Á gómez-Ríos, MD, Principal Investigator — C.H.U. A Coruña
Locations (1):
- Teresa Herrera Hospital; A Coruña University Hospital Complex, A Coruña, A Coruña, Spain

REFERENCES:
- [Background] Moiniche S, Mikkelsen S, Wetterslev J, Dahl JB. A qualitative systematic review of incisional local anaesthesia for postoperative pain relief after abdominal operations. Br J Anaesth. 1998 Sep;81(3):377-83. doi: 10.1093/bja/81.3.377. PMID 9861124
- [Background] Mecklem DW, Humphrey MD, Hicks RW. Efficacy of bupivacaine delivered by wound catheter for post-Caesarean section analgesia. Aust N Z J Obstet Gynaecol. 1995 Nov;35(4):416-21. doi: 10.1111/j.1479-828x.1995.tb02156.x. PMID 8717568
- [Background] Liu SS, Richman JM, Thirlby RC, Wu CL. Efficacy of continuous wound catheters delivering local anesthetic for postoperative analgesia: a quantitative and qualitative systematic review of randomized controlled trials. J Am Coll Surg. 2006 Dec;203(6):914-32. doi: 10.1016/j.jamcollsurg.2006.08.007. Epub 2006 Oct 25. No abstract available. PMID 17116561
- [Background] Lavand'homme PM, Roelants F, Waterloos H, De Kock MF. Postoperative analgesic effects of continuous wound infiltration with diclofenac after elective cesarean delivery. Anesthesiology. 2007 Jun;106(6):1220-5. doi: 10.1097/01.anes.0000267606.17387.1d. PMID 17525598
- [Background] Ranta PO, Ala-Kokko TI, Kukkonen JE, Ohtonen PP, Raudaskoski TH, Reponen PK, Rawal N. Incisional and epidural analgesia after caesarean delivery: a prospective, placebo-controlled, randomised clinical study. Int J Obstet Anesth. 2006 Jul;15(3):189-94. doi: 10.1016/j.ijoa.2006.02.003. PMID 16798442
- [Background] Zohar E, Shapiro A, Eidinov A, Fishman A, Fredman B. Postcesarean analgesia: the efficacy of bupivacaine wound instillation with and without supplemental diclofenac. J Clin Anesth. 2006 Sep;18(6):415-21. doi: 10.1016/j.jclinane.2006.01.001. PMID 16980157
- [Background] Zohar E, Luban I, Zunser I, Shapiro A, Jedeikin R, Fredman B. Patient-controlled bupivacaine wound instillation following cesarean section: the lack of efficacy of adjuvant ketamine. J Clin Anesth. 2002 Nov;14(7):505-11. doi: 10.1016/s0952-8180(02)00422-1. PMID 12477585
- [Background] Bamigboye AA, Hofmeyr GJ. Caesarean section wound infiltration with local anaesthesia for postoperative pain relief - any benefit? S Afr Med J. 2010 May 4;100(5):313-9. doi: 10.7196/samj.3716. PMID 20460027
- [Background] Bamigboye AA, Hofmeyr GJ. Local anaesthetic wound infiltration and abdominal nerves block during caesarean section for postoperative pain relief. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006954. doi: 10.1002/14651858.CD006954.pub2. PMID 19588413
- [Background] Dahl JB, Moiniche S, Kehlet H. Wound infiltration with local anaesthetics for postoperative pain relief. Acta Anaesthesiol Scand. 1994 Jan;38(1):7-14. doi: 10.1111/j.1399-6576.1994.tb03830.x. No abstract available. PMID 8140877
- [Derived] Gomez-Rios MA, Codesido-Barreiro P, Seco-Vilarino C, Calvin-Lamas M, Curt-Nuno F, Nieto-Serradilla L, Rabunal-Alvarez MT, Fernandez-Rodriguez F, Peteiro-Cartelle J, Pensado-Boo R, Bou G, Pensado-Castineiras A, Casans-Frances R. Wound Infusion of 0.35% Levobupivacaine Reduces Mechanical Secondary Hyperalgesia and Opioid Consumption After Cesarean Delivery: A Prospective, Randomized, Triple-Blind, Placebo-Controlled Trial. Anesth Analg. 2022 Apr 1;134(4):791-801. doi: 10.1213/ANE.0000000000005917. PMID 35086112